CLINICAL TRIAL: NCT01712919
Title: IMRT With Concurrent Chemotherapy and Cetuximab Against Locoregionally Advanced NPC: a Phase 1 Study
Brief Title: Chemoradiation Plus Weekly c225 Against Locoregionally Advanced Nasopharyngeal Carcinoma (NPC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu Cancer Institute & Hospital (Other)
Responsible Party: Principal Investigator, Dr. Xia He, Director of the department of radiation oncology, Jiangsu Cancer Institute & Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LA-chemoR-c225; JSCC-SACT-01 (Other: Department of Radiation Oncology,Jiangsu Cancer Hospital)
Record Dates: First submitted 2012-10-18; First posted 2012-10-24 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2014-03

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Locoregionally advanced nasopharyngeal carcinoma; cetuximab; chemoradiation
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Radiotherapy, Intensity-Modulated; Paclitaxel; nedaplatin; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- cetuximab (Experimental): Patients will be given intensity-modulated radiotherapy,2 cycles of concurrent chemotherapy with paclitaxel and nedaplatin,and weekly cetuximab during radiation therapy.
  Interventions: Radiation: Intensity-modulated radiotherapy; Drug: Concurrent chemotherapy with paclitaxel and nedaplatin; Biological: Cetuximab

INTERVENTIONS:
Radiation: Intensity-modulated radiotherapy — Patients will be given intensity-modulated radiotherapy(IMRT)
Drug: Concurrent chemotherapy with paclitaxel and nedaplatin — Patients will be given 2 cycles of concurrent chemotherapy with paclitaxel and nedaplatin
Biological: Cetuximab — Patients will be given cetuximab weekly during radiation therapy

SUMMARY:
The investigators will add weekly cetuximab (c225) to the standard care of chemoradiation against locoregionally advanced Nasopharyngeal Carcinoma (NPC), and evaluate the toxicity and efficacy of this new regimen.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed untreated NPC patients
* locoregionally advanced (T3-4 or N2-3 M0)
* 18-65 years
* with MRI examinations
* ECOG ≤ 2
* With written consent

Exclusion Criteria:

* Without a second cancer
* Pregnancy
* With other severe diseases (blood,liver ,kidney or heart diseases)
* Could not be staged properly
* Without written consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2010-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety | 6 months
Number of Participants with Adverse Events as a Measure of Safety and tolerability | 6 months

SECONDARY OUTCOMES:
Progress free survival | 24 months

OTHER OUTCOMES:
local-relapse free survival | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Xia He, M.D. Ph.D., Principal Investigator — Jiangsu Cancer Institute & Hospital
Locations (1):
- Jiangsu Cancer Hospital, Nanjing, Jiangsu, China